CLINICAL TRIAL: NCT01726374
Title: A Single Group Trial Evaluating One Cycle of Adjuvant BEP Chemotherapy in High Risk, Stage 1 Non-seminomatous Germ Cell Tumours of the Testis (NSGCTT)
Brief Title: Trial of 1 Cycle of Adjuvant BEP Chemotherapy in High Risk, Stage 1 Non-seminomatous Germ Cell Testis Tumours
Acronym: 111
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2008/10019; ISRCTN37875250 (Registry Identifier: ISRCTN); 2008-006295-29 (EudraCT Number); 09/H1102/86 (Other: Main REC); CRUK/09/011 (Other Grant/Funding Number: CRUK)
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Stage I Testicular Non-Seminomatous Germ Cell Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One cycle adjuvant BEP(500) (Experimental): Etoposide 165 mg/m2 IV infusion - days 1, 2, 3 Cisplatin 50 mg/m2 IV infusion - days 1, 2 Bleomycin 30,000 IU IV infusion - days 1 (or 2), 8, 15
  Interventions: Drug: BEP(500)

INTERVENTIONS:
Drug: BEP(500) — One cycle of BEP(500):
  Etoposide 165 mg/m2 IV infusion - days 1, 2, 3 Cisplatin 50 mg/m2 IV infusion - days 1, 2 Bleomycin 30,000 IU IV infusion - days 1 (or 2), 8, 15

SUMMARY:
High-risk stage 1 NSGCTTs are curable with careful surveillance followed by 3 cycles of BEP (bleomycin, etoposide, cisplatin with 500mg/m2 of etoposide per cycle) chemotherapy for the 40-50% of cases experiencing recurrence. Alternatively, adjuvant chemotherapy with 2 cycles of BEP(at a lower dose than that used for advanced disease - etoposide 360mg/m2) for these patients achieves the same outcome and avoids intensive surveillance, but delivers 33% more chemotherapy cycles on a population basis.

If a single cycle of BEP at the dose used in advanced disease had a similar high rate of relapse-free survival (cure) to that seen with two lower dose cycles, this would reduce the overall burden of chemotherapy and healthcare resource usage and would be likely to lead to a change in practice globally.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-seminomatous germ cell tumour of combined GCT (NSGCT + seminoma)of the testis
* Histologically proven vascular invasion of the primary tumour into the testicular veins or lymphatics
* Clinical stage 1 patients (normal AFP and HCG, or optimum marker decline approaching normal levels after orchidectomy AND no evidence of metastases on CT of chest, abdomen and pelvis)
* Men aged 16 years or over
* Creatinine clearance > 50 ml/min
* No previous chemotherapy
* WBC > 1.5 x 10^9/l and platelets 100 x 10^9/l
* Fit to receive chemotherapy
* Able to start BEP(500) chemotherapy as part of 111 study within 6* weeks of orchidectomy
* Written informed consent *If there are unavoidable delays this timescale can be extended to 8 weeks

Exclusion Criteria:

* All patients with pure seminoma
* All patients with non-seminoma or combined NSGCT + seminoma > stage 1
* All patients with no vascular invasion
* Previous chemotherapy
* Patients with second malignancy except contralateral TIN and contralateral germ cell tumour treated by orchidectomy and subsequent surveillance of more than 3 years
* Co-morbidity precluding the safe administration of BEP(500) chemotherapy
* Patients with renal function impairment (bilirubin >1.25 x ULN and/or AST >2 x ULN)
* Patients with pre-existing neuropathy
* Patients with pulmonary fibrosis
* Patients with serious illness or medical conditions incompatible with the protocol

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Recurrence | 2 years
  To demonstrate that one cycle of adjuvant BEP(500) reduces 2 year recurrence rate to less than 5%

SECONDARY OUTCOMES:
Immediate and delayed toxicity including long-term permanent infertility (>2 years) | 0 - > 2 years
Relapse free survival | Patients followed up for 5 years
Overall survival | Patients followed up for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Professor Michael Cullen, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (35):
- United Kingdom (35):
  - Guy's Hospital, London, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Aberdeen Royal Infirmary, Aberdeen
  - Ysbyty Gwynedd, Bangor
  - Queen Elizabeth Hospital, Birmingham
  - Royal Sussex County Hospital, Brighton
  - Bristol Haematology and Oncology Centre, Bristol
  - Queen's Hospital, Burton-on-Trent
  - Addenbrooke's Hospital, Cambridge
  - Cheltenham General Hospital, Cheltenham
  - Gloucestershire Royal Hospital, Cheltenham
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Royal Derby Hospital, Derby
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Castle Hill Hospital, Hull
  - Ipswich Hospital, Ipswich
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Clatterbridge Centre for Oncology, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - Maidstone Hospital, Maidstone
  - James Cook University Hospital, Middlesbrough
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Result] Cullen M, Huddart R, Joffe J, Gardiner D, Maynard L, Hutton P, Mazhar D, Shamash J, Wheater M, White J, Goubar A, Porta N, Witts S, Lewis R, Hall E; 111 Trial Management Group. The 111 Study: A Single-arm, Phase 3 Trial Evaluating One Cycle of Bleomycin, Etoposide, and Cisplatin as Adjuvant Chemotherapy in High-risk, Stage 1 Nonseminomatous or Combined Germ Cell Tumours of the Testis. Eur Urol. 2020 Mar;77(3):344-351. doi: 10.1016/j.eururo.2019.11.022. Epub 2020 Jan 1. PMID 31901440